CLINICAL TRIAL: NCT00625586
Title: A Phase 2 Evaluation of the Monoclonal Antibody, RAV12, in Combination With Standard Gemcitabine in the Treatment of Patients With Metastatic Pancreatic Cancer Who Have Not Been Previously Treated for Metastatic Disease
Brief Title: Monoclonal Antibody RAV12 and Gemcitabine in Treating Patients With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000587562; RAVENBIO-RV12-2007-003 (Other: MacroGenics, Inc.)
Record Dates: First submitted 2008-02-26; First posted 2008-02-28 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAV12 plus gemcitabine (Experimental)
  Interventions: Biological: RAV12; Drug: Gemcitabine

INTERVENTIONS:
Biological: RAV12 — RAV12 at 0.375 mg/kg weekly escalated to 0.75 mg/kg weekly, intravenously.
Drug: Gemcitabine — 1000 mg/m2 weekly, intravenously
  Other Names: Gemzar

SUMMARY:
RATIONALE: Monoclonal antibodies, such as RAV12, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving RAV12 together with gemcitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and best dose of monoclonal antibody RAV12 when given together with gemcitabine in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of monoclonal antibody RAV12 when administered with standard gemcitabine hydrochloride in patients with previously untreated metastatic pancreatic cancer.
* To determine the proportion of these patients surviving at 8 months after initiation of this regimen.
* To provide point estimates for response rate and duration of response in patients treated with this regimen.
* To define the toxicity profile of this drug in these patients when administered with standard gemcitabine hydrochloride.
* To estimate, preliminarily, the progression-free survival and overall survival of these patients after treatment with this regimen.
* To explore the utility of the tumor marker, carbohydrate antigen 19-9 (CA19-9), in the assessment of these patients.

OUTLINE: This is a dose-escalation study of monoclonal antibody RAV12, followed by an efficacy study. The study is conducted in two segments.

* Segment 1 (dose escalation of RAV12): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, and 22 of course 1 and on days 1, 8, and 15 of each subsequent course. Patients also receive RAV12 IV once weekly on days 1, 8, and 15 or twice weekly on days 1, 4 or 5, 8, 11 or 12, 15, and 18 or 19 until the maximum tolerated dose (MTD) is reached. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Segment 2 (efficacy): Once the MTD has been determined, patients receive RAV12 at the MTD and gemcitabine hydrochloride as in segment 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained for pharmacokinetic sampling during the dose-escalation segment of the study. Samples are analyzed to determine plasma concentrations of RAV12, gemcitabine hydrochloride, and difluorodeoxyuridine. Blood samples are also examined periodically for expression of serum biomarkers (i.e., CA19-9, RAAG12, and HACA) and for DNA analysis of Fc-gamma receptor polymorphisms. Archival paraffin blocks or slides from biopsy of primary or metastatic deposit or fresh/frozen tissue may be obtained at baseline for additional correlative studies. Samples are analyzed by immunohistochemistry (IHC) for expression of RAAG12 and for development of a companion RAAG12 diagnostic assay.

After completion of study therapy, patients are followed every 8 weeks for up to 3 years.

PROJECTED ACCRUAL: This study will accrue a total of 18 patients in the dose-escalation segment and 63 patients in the efficacy segment of the trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease

    * No prior therapy for metastatic disease (except prior adjuvant chemotherapy and/or radiotherapy)
* At least 1 radiographically measurable site of disease ≥ 2 cm in the largest dimension by traditional CT technique or ≥ 1 cm by spiral CT scan (per RECIST)
* No known history of current or prior central nervous system (CNS) metastatic disease

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase and γ-glutamyltransferase ≤ 2.5 times ULN
* Amylase and lipase ≤ 1.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* Creatinine < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be available for study-related treatments and assessments at the treating institution
* No known hypersensitivity to any component of gemcitabine hydrochloride
* No known hypersensitivity to murine or recombinant proteins, polysorbate 80, or any excipient contained in the drug formulation
* No other primary malignancy that has been in remission for ≤ 3 years except treated nonmelanoma skin cancer, biopsy-confirmed carcinoma in situ of the cervix, squamous intraepithelial lesion on Papanicolaou smear, localized prostate cancer with Gleason score < 6, or resected melanoma in situ
* No other primary malignancy that has a generally accepted recurrence risk ≥ 10%
* No active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 4 weeks of enrollment
* No history of chronic or recurrent infections that require continuous use of antiviral, antifungal, or antibacterial agents
* No serious underlying medical condition that would impair the patient's ability to receive or tolerate the planned treatment at the investigational site, including significant pulmonary compromise or heart disease of New York Heart Association class III or IV
* No dementia or altered mental status that would preclude sufficient understanding to provide informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior and no other concurrent investigational agents
* More than 1 week since prior oral antiviral, antifungal, or antibacterial therapy
* No concurrent immunosuppressive medications, steroids (except steroid inhaler, ophthalmic solution, nasal spray, or a stable dose of ≤ 10 mg/day of oral prednisone or equivalent), other antineoplastic therapy, or antitumor vaccinations
* Monoclonal antibody treatment for non-cancer indications must be completed at least 3 half lives from study entry
* No concurrent prophylactic hematologic growth factors
* No concurrent megavitamin therapy
* No concurrent bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-04-15; Primary Completion 2009-01-21 (Actual); Study Completion 2009-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanford Stewart, MD, Study Chair — MacroGenics, Incorporated
Locations (2):
- United States (2):
  - MacroGenics, Incorporated, South San Francisco, California
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment was conducted by two cancer institutes between April and July 2008.
Groups:
- RAV12 Plus Gemcitabine: RAV12 monoclonal antibody plus gemcitabine
Period: Overall Study
Arm/Group | RAV12 Plus Gemcitabine
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Groups:
- RAV12 Plus Gemcitabine: Escalating doses of RAV12, plus standard gemcitabine at 1000 mg/m2 iv over 30 min., weekly days 1, 8, 15, 22 of the first cycle and 1000 mg/m2 iv over 30 min., weekly days 1, 8, and 15 of each subsequent cycle of 28 days
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (NA) — Only 2 patients enrolled. Statistical analysis not performed.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients Alive at 12 Months
Time Frame: 12 months
Population: The study was terminated at 11 months. There is no 12 month data.
Groups:
- RAV12 Plus Gemcitabine: RAV12 plus standard gemcitabine
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Partial Response and Complete Response Rates
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.0; partial response = 30% decrease in sum of longest diameter. complete response = 100% decrease in sum of longest diameter. Rate of response = proportion of complete or partial responses based on number of patients evaluated.
Time Frame: 8 months
Population: Only 1 patient was evaluable for response assessment.
Measure: Number; unit: participants
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Median Progression-free Survival
Description: Time from the first dose date to the date of first documented progression or death from any cause, whichever occurs first.
Time Frame: up to 11 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
months | 4.5 (4.94)

4. Secondary Outcome: Median Overall Survival
Description: Time from the first dose date to the date of death from any cause
Time Frame: up to 11 months
Population: Survival data is only available for 1 patient. The second patient was known to be alive at 9 months but lost to follow up. Median overall survival cannot be calculated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
months | NA [NA to NA] — Median overall survival could not be calculated due to an insufficient number of events

5. Secondary Outcome: Participants With Adverse Events
Description: Frequency of adverse events and serious adverse events
Time Frame: Throughout the study, up to 11 months
Measure: Number; unit: participants
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
participants | 2

6. Secondary Outcome: Cmax
Description: RAV12 and gemcitabine cmax
Time Frame: 29 days
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
mcg/mL | NA (NA) — Cmax could not be calculated due to insufficient number of samples

7. Primary Outcome: Number of Patients Alive at 8 Months
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | RAV12 Plus Gemcitabine
Number analyzed (Participants) | 2
participants | 1

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 11 months
Arm/Group | RAV12 Plus Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAV12 Plus Gemcitabine (N=2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Leg pain (General disorders) | 1
Edema (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAV12 Plus Gemcitabine (N=2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (2)
Chest discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (4)
Platelet count decreased (Investigations) | 2 (6)
Urine colour abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No